CLINICAL TRIAL: NCT02947074
Title: Meditation Practice in Pediatric Healthcare Professionals: a Randomized Controlled Clinical Trial
Brief Title: Meditation Practice in Pediatric Healthcare Professionals
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Danilo Forghieri Santaella (Other)
Collaborators: Federal University of São Paulo (Other)
Responsible Party: Sponsor-Investigator, Danilo Forghieri Santaella, Ph.D., University of Sao Paulo
Organization: University of Sao Paulo (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 50822215.9.0000.5505:
Record Dates: First submitted 2016-10-06; First posted 2016-10-27 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Stress, Psychological
Keywords: Yoga; Meditation; Glutathione; Catecholamine; polysomnography
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Waiting list
- Yoga Meditation (Experimental): Previously naive to yoga and meditation, subjects will receive 2 30min yoga meditation classes for 8 weeks.
  Interventions: Behavioral: Yoga Meditation

INTERVENTIONS:
Behavioral: Yoga Meditation — Briefly, subjects will be taught to progressively drive their attention to their inner-self, and keep a calm, nonjudgmental and observational approach towards their own thoughts for 30 minutes.
  Arms: Yoga Meditation

SUMMARY:
Rationale: Healthcare professionals face a growing burden of responsibilities and work overload which may cause psychological suffering expressed by burnout, depression and other negative psychological variables. Personal behavioral strategies may facilitate the coping process. To maintain these positive characteristics, it is necessary that one decouples from automatic thoughts, habits and patterns of unhealthy behaviors, leading to behavioral and physiological regulation, through mindfulness techniques. More specifically, Yoga is an ancient Indian philosophical and practical system and its ultimate goal is to calm the human mind, and increase vital capabilities. In addition to the ethical precepts of Yoga, practices involve asanas (postures), pranayama (breathing exercises) and dhyana (meditation). Many studies have shown the positive effects of Yoga and meditation on psychometric variables, however, there are few which address the effectiveness of Yoga on improving psychometric variables of health care professionals. Thus, aiming to reduce the symptoms that health care professionals experience when they are under burnout, this study intends to use Yoga meditation, which may enable the professional to experience decoupling of harmful feelings, improving, firstly, one's own inner self-relationship and therefore, with patients and their families.

Objective: To investigate the effects of a 8-week yoga meditation program on psychometric and physiological variables of Pediatrics health professionals.

Methods: randomized controlled clinical trial. Participants: 60 health professionals from the Pediatrics Department of a tertiary hospital from Federal University of São Paulo (UNIFESP) will be randomized to meditation or control (waiting list) groups. Subjects of the meditation groups will have 2 30 min classes a week.

Evaluations: Psychometric and physiological variables will be accessed at study entry (baseline) and after its completion (8-weeks).

Statistical Analysis: mixed general linear model (intervenient factors: groups - meditation vs. control and moment - baseline vs. 8-weeks). Significance accepted with p<0.05.

DETAILED DESCRIPTION:
Rationale: Healthcare professionals face a growing burden of responsibilities and work overload which may cause psychological suffering expressed by burnout, depression and other negative psychological variables. On the other hand, there are individual strategies which may be involved and facilitate the coping process: resilience, self-compassion, subjective well-being, subjective quality of life. In order to maintain these positive characteristics, it is necessary that one may decouple from automatic thoughts, habits and patterns of unhealthy behaviors, leading to behavioral and physiological regulation. There are many mindfulness techniques, which hold in common the following operating parameters: use of a specific technique, clearly defined and regularly practiced; use of muscle relaxation during the process; existence of logical relaxation without the intention of analyzing, judging or creating any expectation about the process. Specifically, Yoga is an ancient Indian philosophical and practical system and its ultimate goal is to calm the human mind, and increase vital capabilities. In addition to the ethical precepts of Yoga, its practices involve asanas (postures), pranayama (breathing exercises) and dhyana (meditation). Therefore, the process must be done in a gradual and progressive manner, from the outermost to the innermost, from the simplest to the most complex - from the body to the mind, with breath as a bridge between them. Many studies have shown the positive effects of Yoga and meditation on psychometric variables, however, there are few which address the effectiveness of Yoga on improving psychometric variables of health care professionals. Thus, aiming to reduce the symptoms that health care professionals suffer when they are in burnout, this study intends to use Yoga meditation, which may enable health professionals to experience decoupling of harmful feelings, improving one's own inner self-relationship and therefore, with patients and their families.

Primary Objective: To assess whether a 8-week intervention of a yoga meditation program influences psychometric (burnout, resilience, self-compassion, subjective well-being, health related quality of life and mindfulness) and physiological (polysomnography, glutathione, catecholamine and serotonin) variables of Pediatrics health professionals.

Secondary Objective: To investigate the cross psychometric profile of Federal University of São Paulo (UNIFESP) Pediatrics professionals at the inception of the program.

Methodology Experimental design: randomized controlled clinical trial.

Participants: 60 health professionals from the Pediatrics Department of a tertiary hospital from UNIFESP will be randomized to meditation or control (waiting list) groups. At the end of the protocol participants of the control group will be offered the possibility to participate of an identical meditation program. Inclusion criteria: adults; both sexes; not diagnosed with psychiatric/cognitive disorder or taking any medication which might bias the evaluation process. The intervention group will participate in an 8-week course of meditation (2 30-min classes a week).

Space: Evaluations and meditation program will be conducted in a quiet room specifically reserved for this training at UNIFESP.

Primary outcome: Demonstrate that meditation can be a useful tool in improving burnout, resilience, self-compassion, subjective well-being, quality of life and of health care professionals.

Resources: All personnel and logistics necessary for this research will be provided by the Sports Center of the University of São Paulo (CEPEUSP) and UNIFESP.

Procedures: Meditation training will follow a weekly stratified plan, through which participants will be guided from the most exterior perceptions, towards the inner most ones, focusing on yoga meditation processes. First week will have relaxation, and easy-to-perform asanas along with introduction to pranayama; second week will have pranayamas and introduction to concentration; from third week onwards, participants will have concentration and meditation as main components of the classes.

Evaluation plan: Measurements will be done in two stages: study entry and after 8 weeks. Assessment instruments: burnout (MBI-HSS), resilience (BRCS), self-pity (SCS), subjective well-being (EBE), quality of life (WHOQOL BREF), attention and mindfulness (MAAS) scales; venous puncture (by a nurse from Clinical Studies Development Centre Brazil) - 20ml of blood for glutathione, catecholamine and serotonin analysis; polysomnography (Sleep Institute - São Paulo, Brazil).

Statistical Analysis: mixed general linear model (intervenient factors: groups - meditation vs. control and moment - baseline vs. 8-weeks). Significance accepted with p<0.05.

Potential impact: Investigators expect to have a great positive impact on health care professionals. Through meditation, participants may improve burnout rates, resilience, self-compassion, subjective well-being, quality of life and mindfulness. Such improvements may improve work environment, work satisfaction, decrease absenteeism and increase the professional-patient relationship. Besides, with positive results, it is possible to try and spread the practice of Yoga to other public hospitals.

ELIGIBILITY:
Inclusion Criteria:

* adults
* both genders
* naive to yoga
* naive to meditation

Exclusion Criteria:

* diagnosed with psychiatric/cognitive disorder
* taking any medication which might bias the evaluation process
* illiterate.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-07; Primary Completion 2017-12 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Change in Glutathione from baseline to 8 weeks | Baseline and 8-weeks
  Spectrometry

SECONDARY OUTCOMES:
Change in Catecholamines from baseline to 8 weeks | Baseline and 8-weeks
  HPLC
Change in Serotonin from baseline to 8 weeks | Baseline and 8-weeks
  Elisa
Change in Burnout from baseline to 8 weeks | Baseline and 8-weeks
  MBI-HSS
Change in Resilience from baseline to 8 weeks | Baseline and 8-weeks
  BRCS
Change in Self-compassion from baseline to 8 weeks | Baseline and 8-weeks
  SCS
Change in Subjective well-being from baseline to 8 weeks | Baseline and 8-weeks
  EBE
Change in Quality of life from baseline to 8 weeks | Baseline and 8-weeks
  WHOQOL - BREF
Change in Mindfulness from baseline to 8 weeks | Baseline and 8-weeks
  MAAS

CONTACTS AND LOCATIONS:
Overall Officials: Priscilla C Guerra, Master, Principal Investigator — Federal University of São Paulo
Locations (1):
- UNIFESP, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moss M, Good VS, Gozal D, Kleinpell R, Sessler CN. An Official Critical Care Societies Collaborative Statement-Burnout Syndrome in Critical Care Health-care Professionals: A Call for Action. Chest. 2016 Jul;150(1):17-26. doi: 10.1016/j.chest.2016.02.649. PMID 27396776
- [Background] Blackwelder R, Watson KH, Freedy JR. Physician Wellness Across the Professional Spectrum. Prim Care. 2016 Jun;43(2):355-61. doi: 10.1016/j.pop.2016.01.004. PMID 27262013
- [Background] Cardoso R, de Souza E, Camano L, Leite JR. Meditation in health: an operational definition. Brain Res Brain Res Protoc. 2004 Nov;14(1):58-60. doi: 10.1016/j.brainresprot.2004.09.002. PMID 15519952
- [Background] Tang YY, Posner MI. Tools of the trade: theory and method in mindfulness neuroscience. Soc Cogn Affect Neurosci. 2013 Jan;8(1):118-20. doi: 10.1093/scan/nss112. Epub 2012 Oct 18. PMID 23081977
- [Background] Travis F, Shear J. Focused attention, open monitoring and automatic self-transcending: Categories to organize meditations from Vedic, Buddhist and Chinese traditions. Conscious Cogn. 2010 Dec;19(4):1110-8. doi: 10.1016/j.concog.2010.01.007. Epub 2010 Feb 18. PMID 20167507
- [Background] Chiesa A, Malinowski P. Mindfulness-based approaches: are they all the same? J Clin Psychol. 2011 Apr;67(4):404-24. doi: 10.1002/jclp.20776. Epub 2011 Jan 19. PMID 21254062
- [Background] Goyal M, Singh S, Sibinga EM, Gould NF, Rowland-Seymour A, Sharma R, Berger Z, Sleicher D, Maron DD, Shihab HM, Ranasinghe PD, Linn S, Saha S, Bass EB, Haythornthwaite JA. Meditation programs for psychological stress and well-being: a systematic review and meta-analysis. JAMA Intern Med. 2014 Mar;174(3):357-68. doi: 10.1001/jamainternmed.2013.13018. PMID 24395196
- [Background] Barnes PM, Bloom B, Nahin RL. Complementary and alternative medicine use among adults and children: United States, 2007. Natl Health Stat Report. 2008 Dec 10;(12):1-23. PMID 19361005
- [Background] Pastori D, Pignatelli P, Farcomeni A, Menichelli D, Nocella C, Carnevale R, Violi F. Aging-Related Decline of Glutathione Peroxidase 3 and Risk of Cardiovascular Events in Patients With Atrial Fibrillation. J Am Heart Assoc. 2016 Sep 8;5(9):e003682. doi: 10.1161/JAHA.116.003682. PMID 27609361
- [Derived] Guerra PC, Santaella DF, D'Almeida V, Santos-Silva R, Tufik S, Len CA. Yogic meditation improves objective and subjective sleep quality of healthcare professionals. Complement Ther Clin Pract. 2020 Aug;40:101204. doi: 10.1016/j.ctcp.2020.101204. Epub 2020 May 30. PMID 32891281